CLINICAL TRIAL: NCT03541330
Title: Information and Accompaniment of Siblings Following the Announcement of a Cancer in Pediatric Hematology.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: default of inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016_83; 2016-A02091-50 (Other: ID-RCB Number, ANSM)
Record Dates: First submitted 2017-03-08; First posted 2018-05-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Malignant Haemopathy
Keywords: Siblings; information; malignant haemopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- siblings (Other): Brother or sister of a child has malignant haemopathy and follow-up in the pediatric hematology department
  Interventions: Other: semi-directive interview

INTERVENTIONS:
Other: semi-directive interview — semi-structured interview conducted by a clinical psychologist

SUMMARY:
The primary objective is to evaluate the experience with the information received on the disease by the healthy brothers and sisters of childrens with malignant haemopathy at the Centre Hospitalier Régional et Universitaire of Lille

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 12 years old
* Brother or sister of a child:

O has malignant haemopathy O follow-up in the pediatric hematology department in Lille, O diagnosed from 6 weeks to 1 year before maintenance of the healthy subject included

* whose parents are able to understand and sign voluntarily informed consent
* Affiliated to a social security scheme
* Ability to understand and answer questions alone during the semi-structured interview

Exclusion Criteria:

* Child under 6 years or over 12 years
* Subject with a pathology that may interfere with the course of the study, according to the investigator's assessment
* Absence of the informed consent of one of the parents and / or the legal representative
* Refusal of participation of the subject

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Level of satisfaction and characteristics of information received about the disease by healthy siblings of children with hematological malignancies | 1 year
  Measure Qualitative Interviews by Grounded theory. The experience with the information received on the disease by the healthy brothers and sisters of childrens with malignant haemopathy.
  Assessment of the level of satisfaction with the information received. The information will be characterized according to three dimensions: the framework (by whom, with whom, where, when, how) and the content of the information

SECONDARY OUTCOMES:
Explore the representations of the disease in healthy siblings | 1 year
  The representation of the disease is the set of personal beliefs of an individual about the disease. It allows him to make sense of the disease. These data will be analyzed during the semi-structured interview
Evaluate their information and support needs following the announcement of the disease | 1 year
  information and support needs gathered during the semi-structured interview
Identify the possible psychic and social consequences of the disease in these healthy subjects | 1 year
  to identify during the semi-directive interview the elements informing about the social behavior and the psychic state of the subject included, expressed spontaneously by the subject, directly (in the speech, for example "I am sad") or indirectly (by attitude, for example: crying)

CONTACTS AND LOCATIONS:
Overall Officials: Eva De Berranger, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No